CLINICAL TRIAL: NCT04723524
Title: Multi-center, Randomized, Double Blind and Placebo Controlled Clinical Trial on the Effectiveness and Safety of Jinhua Qinggan Granules (JHQG) for the Treatment of COVID 19 Patients
Brief Title: Jinhua Qinggan Granules in the Treatment of COVID-19
Acronym: RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Indus Hospital and Health Network (Other); Dow University Hospital, Mission Rd, Gulzar-e-Hijri, Scheme 33, Karachi. Tel: (92-21) 38771111 (Unknown); Dr. Ruth K.M. Pfau Civil Hospital, Karachi (Other Government)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-003-TCM- JHQG -2020/3.0
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — jinhua qinggan granules; Medicine, Chinese Traditional

STUDY DESIGN:
Intervention Model Description: Multi-center, Randomized, Double Blind and Placebo Controlled Clinical Trial
Who Masked: Participant, Care Provider
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): 150 Cases, treated with Jinhua Qinggan (JHQG) Granules
  Interventions: Combination Product: Jinhua Qinggan (JHQG) Granules, Traditional Chinese Medicine
- Control group (Placebo Comparator): 150 Cases, Placebo treated
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Combination Product: Jinhua Qinggan (JHQG) Granules, Traditional Chinese Medicine — Jinhua Qinggan granules: 5g/sachet; 1 sachet each time, 3 times daily after meal, dissolve in boil water.
  Arms: Treatment group
Other: Placebo Comparator — Jinhua Qinggan granules simulation (placebo) agent: 5g/sachet; 1 sachet each time, 3 times daily after meal, dissolve in boil water.
  Arms: Control group

SUMMARY:
The clinical trial is designed to be randomized, double blind, placebo controlled, to evaluate the effectiveness and safety of Jinhua Qinggan granules (JHQG) on mild-category patients of COVID-19 in Pakistani population with the age limit of 18-75 years, at10th day comprehensive follow-up. The informed consent form must be signed by the subjects before their participation in the trial.

DETAILED DESCRIPTION:
The course of treatment is 10 days, and the visit points are set on the 1st and 10th day, in which 10th day is follow-up. Patients will be assessed by using seven-category ordinal scale and clinical signs and symptoms on 1st and 10th day. If the subject recovers and checks out within 10 days, they will be recorded once before checking out. All effectiveness and safety inspection items will be done once before the trial and once at follow-up point i.e. 10th day. In case of any new abnormality or abnormality aggravation after the treatment, should be followed up until normal or stable.

ELIGIBILITY:
Inclusion Criteria:

* 1) Between the ages of 18-75 years, both male and female.
* 2) Confirmed Coronavirus infection by real time RT-PCR.
* 3) Mild cases of Coronavirus having main symptoms with minimum 2 grade (as mentioned in 7.1.6).
* 4) The subject has signed the informed consent form;

Exclusion Criteria:

* 1) Younger than 18 years or older than 75 years.
* 2) Patients with moderate or critical Coronavirus infection confirmed by real time RT-PCR; cases meeting any of the following criteria:

  1. Lung lesions
  2. Respiratory failure and requiring mechanical ventilation
  3. Shock
  4. With other organ failure that requires ICU cares.
* 3) Severe primary health conditions associated with cardiovascular, cerebrovascular, pulmonary, hepatic, renal, endocrine and hematological diseases, hematopoietic system (above grade II of cardiac function; ALT & AST are 1.5 times higher than the normal value; Creatinine above the upper limit of normal value) and mental illness or serious diseases affecting their survival, such as cancer or AIDS;
* 4) With severe cardiopulmonary dysfunction, cardiopulmonary insufficiency.
* 5) Subjects, who took other antiviral, antibacterial, cough relieving, expectorant and antiasthmatic drugs within 3 days prior to the visit (including β2 receptor agonists, anticholinergic agents, theophylline drugs, glucocorticoids, expectorant and Chinese Medicine.)
* 6) Allergic individuals and those who are known to be allergic to experimental drugs
* 7) Pregnant women, lactating women or fertile women who are ready to conceive in 3 months.
* 8) Subject, who has participated in the past 1 month in another clinical study.
* 9) Subjects who are not suitable for the clinical trial based on investigators' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Change in Primary symptom (cough) | 10th day of treatment.
  A grading symptom from 0-6 will be used to assess the symptom (Cough) where the score will be 0 for No cough, 2 for Intermittent cough, 4 for Cough mildly impacting the daily work and 6 Frequent cough or paroxysmal cough seriously impacting the work and life.
Change in Primary symptom (Fever) | 10th day of treatment
  A grading symptom from 0-6 will be used to assess the improvement of main clinical symptom (Fever) where the score will be 0 for No fever ≤ 37 °C (98.6°F), 2 for body temperature > 37°C (98.6°F) to ≤ 38°C (100.4°F), 4 for body temperature > 38°C (100.4°F) to ≤ 39°C (102.2°F) and 6 for body temperature > 39°C (102.2°F) to ≤ 40°C (104°F).
Time for Negative COVID-19 Test | 2nd follow-up on 10th day or 3rd follow-up for RT-PCR test on 15th day if positive on 10th day
  time for Negative coronavirus (COVID-19) Test on RT-PCR

SECONDARY OUTCOMES:
Body temperature | 10 days
  The onset time of fever and the complete time of defervescence.
white blood cells count | during the 10-day course of treatment
  Change in white blood cells count
C-reactive protein test | during the 10-day course of treatment
  Change in C-reactive protein level in blood
ferritin test | during the 10-day course of treatment
  Change in ferritin level in blood
Radiology | during the 10-day course of treatment
  Change in radiographic findings of the lungs.
Quality of life assessment: | during the 10-day course of treatment
  The quality of life of the product will be assessed by using the Patient's Quality of Life Assessment Questionnaire (QOL). The QOL questionnaire is divided into three parts: Psychology, Physiology, and Society. The score of each section is calculated by the sum of score of the part divided by the number of questions. The total is the sum of the three parts, and the minimum importance difference (MID) is 1.3, which means that if the QOL questionnaire score before and after treatment in the same patient rises by 1.3, it indicates that the treatment is effective. At the same time, the higher the QOL score, the lighter the illness is.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Raza Shah, Principal Investigator — CBSCR , ICCBS, University of Karachi
Locations (1):
- Center for Bioequivalence Studies and Clinical Research (CBSCR), ICCBS, university of Karachi, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Q, Cao F, Wang Y, Xu X, Sun Y, Li J, Qi X, Sun S, Ji G, Song B. The efficacy and safety of Jinhua Qinggan granule (JHQG) in the treatment of coronavirus disease 2019 (COVID-19): A protocol for systematic review and meta analysis. Medicine (Baltimore). 2020 Jun 12;99(24):e20531. doi: 10.1097/MD.0000000000020531. PMID 32541475
- [Derived] Shah MR, Fatima S, Khan SN, Ullah S, Himani G, Wan K, Lin T, Lau JYN, Liu Q, Lam DSC. Jinhua Qinggan granules for non-hospitalized COVID-19 patients: A double-blind, placebo-controlled, and randomized controlled trial. Front Med (Lausanne). 2022 Aug 1;9:928468. doi: 10.3389/fmed.2022.928468. eCollection 2022. PMID 35979216
- See also: The efficacy and safety of Jinhua Qinggan granule (JHQG) in the treatment of coronavirus disease 2019 (COVID-19): A protocol for systematic review and meta analysis. Medicine (Baltimore) — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7302627/